CLINICAL TRIAL: NCT06208566
Title: A Randomized Controlled Trial of a Bot-based Self-help Program (WELL)
Brief Title: A Bot-based Self-help Program (WELL)
Acronym: WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Klagenfurt (Other)
Collaborators: Meta Platforms, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 101095530
Record Dates: First submitted 2023-12-13; First posted 2024-01-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Well-Being, Psychological
Keywords: well-being; digital intervention; randomized trial; conversational agent
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversational Agent Zenny (Experimental): Participants received access to a self-help program delivered via an automated conversational agent on WhatsApp.
  Interventions: Behavioral: Conversational Agent Zenny
- Web-based Wellness Resources (Active Comparator): Participants received a list of three freely accessible wellness resources available on the web.
  Interventions: Behavioral: Web-based Wellness Resources

INTERVENTIONS:
Behavioral: Conversational Agent Zenny — The intervention group involves a newly developed conversational agent self-care program. This program consists of 40 separate modules based on empirically supported techniques. Modules include the following core sections: cognitive behavioral skills, interpersonal relationships, positive psychological growth, relaxation, goal setting, and emotional regulation skills. The modules focus on cognitive-behavioral skills for reducing emotional distress, improving behavioral activation and healthy behaviors, and problem-solving skills. The intervention was delivered via a decision-tree based conversational agent in WhatsApp messenger.
  Arms: Conversational Agent Zenny
Behavioral: Web-based Wellness Resources — The control group involved referral to a menu of freely-available evidence-based wellness resources linked from the study website, "Your Healthiest Self: Wellness Toolkits", "Doing What Matters in Times of Stress", and "How Right Now". These website choices involved self-selection of relevant modules for improving mood, reducing stress and anxiety, addressing relationship problems, and other wellness topics. These programs required only access to the websites and could be completed in a self-help format by participants at their own pace.
  Arms: Web-based Wellness Resources

SUMMARY:
In the current project, the effectiveness of a new bot-based universal prevention program aimed at improving well-being will be developed and tested. This prevention program includes a variety of modules that target common areas related to well-being including interpersonal relationships, emotional regulation, beliefs and behaviors, problem-solving, sleep hygiene, goal setting, personal growth, and healthy habits.

DETAILED DESCRIPTION:
The purpose of the data collection is to evaluate a new intervention as part of a research study.

In the current project, a new bot-based universal prevention program aimed at improving well-being will be developed and tested. This prevention program includes a variety of modules that target common areas related to well-being including interpersonal relationships, emotional regulation, beliefs and behaviors, problem-solving, sleep hygiene, goal setting, personal growth, and healthy habits. The intervention modules are based on existing empirically supported intervention techniques from traditional cognitive-behavioral therapies and other third generation therapies such as mindfulness training and dialectical behavioral therapy. The focus of the program is to introduce psychological concepts that have been shown to be effective for managing emotions and problems to a broader public audience. Another focus is on helping individuals connect with resources that are available related to subjective well-being. Often individuals who may be interested in self-help interventions do not know where to seek help and interventions that they may find (e.g., apps), may not be scientifically valid. By providing recommendations on resources that are specific to an individual's needs, this may reduce one barrier to care.

The focus of this project is not only on testing the effectiveness of the program on well-being compared to an online control condition in a randomized controlled trial, but on improving REACH to individuals who may benefit from such an intervention. Thus, the focus is on brief, low burden assessments, rather than a full battery typical in psychological studies, to improve acceptability, recruitment rates, and retention rates. The implementation science model, RE-AIM, will be used as a framework for this study (http://www.re-aim.org/).

H1: The intervention group will evidence significant improvements in well-being at the post-assessment and follow-up assessments (1-month, 6- month, 12-month) compared to the control group.

H2: The effectiveness of the intervention will be similar across gender and age after controlling for participation/engagement and user satisfaction.

H3: The intervention group will have significantly higher psychological growth compared to the control group at post-assessment and follow-ups assessments (1-month, 6- month, 12-month).

H4: The intervention group will have higher response rates, higher retention rates, and more self-reported active participation/engagement than the control group.

H5: Higher user satisfaction and more active participation/engagement will be associated with greater improvements in well-being.

H6: Higher user satisfaction will lead to subsequent increases in participation/engagement over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* proficient in spoken and written English
* residents of the United States
* provided consent to be eligible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1595 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Subjective well-being | At pre-assessment and 1, 6 and 12 months after pre-assessment
  The WHO-5 Well-Being Scale (WHO-5) is a 5-item short self-reported measure of current subjective wellbeing. Participants are asked to rate the frequency of well-being past month (e.g., "My daily life has been filled with things that interest me") based on a Likert scale from 0 to 5 ("At no time" to "All of the time"). Scores range from 0 to 25 with higher scores indicating higher subjective well-being.
Psychosocial flourishing | At pre-assessment and 1, 6 and 12 months after pre-assessment
  The Flourishing Scale (FS) is an 8-item scale of positive human functioning. Items assess features of human flourishing such as positive relationships, feelings of competence, meaning and purpose in life, and engagement with daily activities. Statements are rated on a 7-point scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Scores can range from 8 to 56, with higher scores reflecting higher well-being.
Psychological well-being | At pre-assessment and 1, 6 and 12 months after pre-assessment
  The Mental Health Continuum Short Form (MHC-SF) measures positive psychological health and comprises 14 items, representing various feelings of well-being. Three items were chosen (happy, interested in life, and satisfied) to represent emotional well-being, six items (one item from each of the 6 dimensions) were chosen to represent psychological well-being, and five items (one item from each of the 5 dimensions) were chosen to represent social well-being. Respondents rate the frequency of every feeling in the past month on a 6-point Likert scale, ranging from 1 (never) to 6 (every day).

SECONDARY OUTCOMES:
User satisfaction | 1 month after pre-assessment
  This is assessed with four items during the post-assessment for both conditions. Satisfaction with the program is formed by individual items on satisfaction, usefulness, relevance, and helpfulness. Participants rate these dimensions on 4-point Likert scales between 0 (strong disagreement) to 4 (strong agreement). Only the item on usefulness is rated on a 5-point Likert scale. A sum score is calculated by summarizing all single item scores, resulting in a range from 0 to 17. Higher scores indicate greater satisfaction with the content.
Participation/Engagement | 1 month after pre-assessment
  This is assessed by the reported frequency using the intervention or control condition resources at the post-assessment. For the first item, participants rate on a 6-point Likert scale how often they participated in the last month, ranged from "not at all" (1) to "daily" (6). On a second item, participants are asked to rate their perceived level of activity on a 4-point Likert scale, ranging from "not at all active" (1) to "very active" (4). The scores for both items are summarized into a sum score, with higher scores indicating greater participation/engagement.

OTHER OUTCOMES:
Module rating of user satisfaction | 1 month after pre-assessment
  Within the intervention group, user satisfaction is assessed following each module. Users are able to rate satisfaction with each completed module from 1 "not at all" (1) to "extremely" (5). An average satisfaction rating across modules over a thirty-day period is computed.
Days chatted bot | 1 month after pre-assessment
  Engagement with the conversational agent is defined as the count of days that a user engaged in conversations within the last 30 days from 0 days to 30 days.
Total messages | 1 month after pre-assessment
  The number of messages sent by the user to the conversational agent is quantified as a further objective measure. This refers to any situation where the user is starting an interaction with the conversational agent or is responding to a message from the conversational agent within the last 30 days from 0 days to 30 days.
Modules started | 1 month after pre-assessment
  This is the total number of modules that is initiated by the participant within the first 30 days, whether they were completed or not (i.e., sum of finished and unfinished modules).
Modules completed | 1 month after pre-assessment
  This is the number of modules that is completed within the first 30 days (i.e., finished modules).
Modules started not completed | 1 month after pre-assessment
  This is the number of modules that is started but not completed within the first 30 days (i.e., unfinished modules).

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Heather, Ph.D., Principal Investigator — University of Klagenfurt; Y-Lan Boureau, Ph.D., Principal Investigator — Meta Platforms
Locations (1):
- Meta Platforms Inc., Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foran HM, Kubb C, Mueller J, Poff S, Ung M, Li M, Smith EM, Akinyemi A, Kambadur M, Waller F, Graf M, Boureau YL. An Automated Conversational Agent Self-Help Program: Randomized Controlled Trial. J Med Internet Res. 2024 Dec 6;26:e53829. doi: 10.2196/53829. PMID 39641985
- See also: Open Science Framework Preregistration (June 3, 2022) — https://archive.org/details/osf-registrations-ahe2r-v1
- See also: Study Website — https://wellsurvey.aau.at/well/project.html